CLINICAL TRIAL: NCT06786650
Title: Comparision of the Analgesic Effects of Intravenous Ibuprofen and Tenoxicam in Acute Migraine Attack
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sinem Dogruyol, Associate Professor Doctor, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-KAEK-18
Record Dates: First submitted 2024-11-29; First posted 2025-01-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Analgesic Affect; Emergency Medicine
Keywords: Anti-Inflammatory Agents Non-Steroidal; Acute migrane attack
MeSH Terms: conditions — Migraine Disorders | interventions — tenoxicam; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Medical treatments will be administered in 100 cc saline to ensure blindness in both treatment groups. The treatment will be prepared by the responsible investigator and will be numbered with the number on the sealed envelope. Thus, it will be ensured that the administering personnel and the patient will be blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenoxicam Group. IV Tenoxicam (Active Comparator): Intravenous tenoxicam (20 mg) will be administered in 100 cc saline in 10 minutes to patients admitted to our emergency department with headache due to acute migraine attack.
  Interventions: Drug: Tenoxicam Injectable Product
- Ibuprofen Group. IV Ibuprofen (Sham Comparator): Intravenous ibuprofen (400 mg) will be administered in 100 cc saline in 10 minutes to patients who present to our emergency department due to headache due to acute migraine attack.
  Interventions: Drug: ibuprofen

INTERVENTIONS:
Drug: Tenoxicam Injectable Product — Analgesic efficacy of the two active agents analysed in our study in acute migraine attack has not been compared before.
  Other Names: tenoxicam
  Arms: Tenoxicam Group. IV Tenoxicam
Drug: ibuprofen — Analgesic efficacy of the two active agents analysed in our study in acute migraine attack has not been compared before.
  Arms: Ibuprofen Group. IV Ibuprofen

SUMMARY:
The aim of this clinical trial is to compare the efficacy of two different non-steroidal anti-inflammatory analgesic drugs in the palliation of headache in acute migraine attack. The main questions it aims to answer are:

1. Is there a difference between the efficacy of two different nonsteroidal anti-inflammatory analgesics?
2. Is there a significant difference between the side effects of two different nonsteroidal anti-inflammatory drugs? Researchers will compare intravenous tenoxicam to intravenous ibuprofen to see if tenoxicam works to treat migraine attack.

Treatments will;

1. be administered in 100 cc saline to ensure blinding in the group.
2. Randomisation will be done by closed envelope method.
3. Numerical Pain Scale (NRS) will be used to evaluate the analgesic efficacy of the drugs. NRS scores will be recorded in both groups before starting treatment (baseline) and at 30, 60 and 120 minutes after treatment.
4. Any side effects due to medication will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65.
* Having a known diagnosis of migraine.
* Exclusion of secondary causes to explain the headache in the emergency department.
* Having migraine during a migraine attack and not having received any medical treatment for migraine before the application.

Exclusion Criteria:

* Being under 18 years of age.
* Being pregnant or breastfeeding.
* Being admitted to the emergency department with headache due to causes other than migraine (secondary).
* Being admitted with an acute migraine attack and having used medication for migraine treatment within 12 hours before admission.
* Having a history of allergy to any of the drugs to be used in the study.
* Having a history of comorbidities for which the drugs to be used in the study are contraindicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Achievement of pain palliation | NRS scores of both patient groups will be recorded at the time of admission (NRS Baseline) and at 30, 60 and 120 minutes after the treatment is given.
  The primary outcome of our study is the achievement of pain palliation. This will be defined as a ≥ 50% reduction in Numerical rating scale (NRS) scores after treatment compared to the baseline score (NRS Baseline). The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Mean and proportional reduction in NRS scores will also be analysed while evaluating the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Colak, Professor Dr, Principal Investigator
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: 12 months ( 01.01.2025-01.01.2026)
Access Criteria: The researcher responsible for data analysis will be authorised to access IPD for 1 year.